CLINICAL TRIAL: NCT01431885
Title: Randomized Controlled Trial of Two Methods of Diagnosing Preterm Labor
Brief Title: Two Methods of Diagnosing Preterm Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010010
Record Dates: First submitted 2011-08-24; First posted 2011-09-12 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Preterm Labor; Preterm Delivery
Keywords: fibronectin; cervical length
MeSH Terms: conditions — Obstetric Labor, Premature; Premature Birth | interventions — Fibronectins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PLAT (Active Comparator): Diagnosis of preterm labor will be made by the March of Dimes Preterm Labor Assessment Toolkit Algorithm B, incorporating transvaginal ultrasound measurement of cervical length, and vaginal fetal fibronectin
  Interventions: Procedure: Diagnosis by cervical length and fibronectin
- Cervical Change (Placebo Comparator): Diagnosis of preterm labor will be made by cervical change by digital examination
  Interventions: Procedure: Cervical change

INTERVENTIONS:
Procedure: Diagnosis by cervical length and fibronectin — Diagnosis will be made by MOD Algorithm B
  Other Names: March of Dimes Preterm Labor Assessment Toolkit Algorithm B
  Arms: PLAT
Procedure: Cervical change — Diagnosis will be made by digital examination of cervical change
  Other Names: None applicable
  Arms: Cervical Change

SUMMARY:
Use of modern diagnostic tools e.g. fetal fibronectin and ultrasound measurement of cervical length to diagnose preterm labor can result in improved outcomes compared to traditional diagnosis based on digital examination to measure cervical change.

DETAILED DESCRIPTION:
Symptomatic preterm labor patients will be randomized to diagnosis of preterm labor by serial digital examination versus an algorithm incorporating transvaginal ultrasound measurement of cervical length and vaginal fetal fibronectin.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic complaints suggestive of preterm labor
* greater than 6 contractions per hour

Exclusion Criteria:

* multiple gestation
* rupture of amniotic membranes
* chorioamnionitis
* congenital malformations
* persistent vaginal bleeding
* abruptio placentae
* placenta previa
* previously diagnosed short cervix < 2.5 cm
* cervical dilation > 3 cm
* cervical cerclage
* exposure to tocolytic drugs
* allergy or contraindication to nifedipine

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2011-08; Primary Completion 2015-02-13 (Actual); Study Completion 2015-02-13 (Actual)

PRIMARY OUTCOMES:
Delivery prior to 37 weeks' gestation | No longer than 18 weeks post randomization (at which time a pregnancy randomized at the earliest possible gestational age would be 42 weeks, generally the contemporary upper limit of the duration of pregnancy)
  Delivery of the baby prior to 37 weeks' gestation by any means and for any reason including spontaneous or indicated delivery for maternal or fetal complications

CONTACTS AND LOCATIONS:
Overall Officials: Conrad R Chao, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Community Regional Medical Center, Fresno, California, United States